CLINICAL TRIAL: NCT05823584
Title: Cell-free DNA From the Junction of Hepatitis B Virus Integration in HCC Patients for Monitoring Post-resection Recurrence: A Comparison Study With Current Biomarkers
Brief Title: Cell-free DNA From Junction of Hepatitis B Virus Integration in HCC Patients for Monitoring Post-resection Recurrence
Status: Completed | Type: Observational
Sponsor: TCM Biotech International Corp. (Industry)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ctDNA-HCC-01
Record Dates: First submitted 2023-04-10; First posted 2023-04-21 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2023-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Hepatitis b Virus; Biomarker; Cell-free DNA; cfDNA; Circulating tumor DNA; ctDNA; virus-host chimera DNA; Chimera DNA
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma、Tissue、ctDNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
HBV DNA integration has been found in the chromosomes of about 90% of HBV-related HCC and the integration site is unique to individual HCC. The virus-host chimera DNA (vh-DNA) from HBV integration sites in HCC a reliable evidence even in the patient with a tiny tumor which is not large enough to be detected by the image scan.

The goal of this observational study is to compare the prediction ability of vh-DNA with the other biomarkers for monitoring the recurrent of HBV-related HCC. The main questions that aim to answer are the sensitivity and specificity of vh-DNA/AFP/ALP-L3/PIVKA-II/TERTC2280 when the gold standard is the guideline of HCC diagnosis.

The surgical tissues and plasma samples from the participants would be collected undergoing the HCC recession surgery when joining the study at the beginning, in order to identify the HBV integration in tumor by Capture NGS and quantify the specific vh-DNA in plasma by ddPCR as personalized biomarkers for minimal residual disease (MRD) monitoring. Moreover, the consistency of vh-DNA from tumor will be validated by pre-operative plasma.

Then the participants will be asked to performed the visit at 2, 5, 8, 11, 14 months after the HCC recession surgery. The plasma sample for vh-DNA/AFP/ AFP-L3/ PIVKA-II/ TERTp C228T testing and the image data from ultrasound, CT or MRI would also be collected at these visits. When the vh-DNA testing result is positive and there is no recurrence at 14 months after the HCC recession surgery, some participants will be asked to followed at 17, 20 months.

Researcher will compare the sensitivity, specificity and predict day of vh-DNA with AFP/ AFP-L3/ PIVKA-II/ TERTp C228T as a biomarker for HCC surveillance. The true value of this novel HBV chimera vh-DNA will be revealed. The results will also support to use for monitoring post-operative recurrence.

In addition, the investigators will explore the performance of TERTp C228T mutation from non-HBV HCC patients. As a different target of ctDNA for HCC, TERTp C228T will be identified using surgical tissues from HCC patients, and plasma samples from the same patient before/after operation will be tested by ddPCR . It will be evaluated that TERTp C228T is predictive or not for recurrence monitoring of HCC.

ELIGIBILITY:
Inclusion Criteria:

1. ≥20 years old.
2. Subject who is diagnosed with HCC
3. Subject who is scheduled to undergo hepatic resection or liver transplant.

Exclusion Criteria:

1. Subject who should not treat with the contrast media (for imaging)
2. Active malignancy (still under intensive cancer treatment or considered in progression) or disease free interval less than one year before entering the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with HCC are scheduled to undergo hepatic resection or liver transplant.
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2019-12-22 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity (vh-DNA vs AFP) (the vh-DNA which could be detected in the pre-operative plasma of participants.) | HCC recurrence within 14 months of post-operative.
  Compare the sensitivity of vh-DNA with AFP as a biomarker for HCC surveillance.

SECONDARY OUTCOMES:
Sensitivity (vh-DNA vs AFP) (the vh-DNA which could not be detected in the pre-operative plasma of participants.) | HCC recurrence within 14 months of post-operative.
  Compare the sensitivity of vh-DNA with AFP as a biomarker for HCC surveillance.
Sensitivity (vh-DNA vs AFP-L3/PIVKA-II/TERTp C228T) | HCC recurrence within 14 months of post-operative.
  Compare the sensitivity of vh-DNA with AFP-L3/ PIVKA-II/ TERTp C228T as a biomarker for HCC surveillance.
Specificity (vh-DNA vs AFP/AFP-L3/PIVKA-II/TERTp C228T) | The 14 months of post-operative.
  Compare the specificity of vh-DNA with AFP/ AFP-L3/ PIVKA-II/ TERTp C228T as a biomarker for HCC surveillance.
Predicted days (vh-DNA vs AFP/AFP-L3/PIVKA-II/TERTp C228T) | HCC recurrence within 14 months of post-operative.
  Compare the predicted day of vh-DNA with AFP/AFP-L3/PIVKA-II/TERTp C228T as a biomarker before HCC recurrence.
Clonality | HCC recurrence within 14 months of post-operative.
  To clarify the clonality of recurrent HCC is same as the original one or is a de novo one.
Sensitivity (TERT C228T vs AFP/AFP-L3/PIVKA-II) | HCC recurrence within 14 months of post-operative.
  Compare the sensitivity of TERTp C228T with AFP/ AFP-L3/ PIVKA-II as a biomarker for HCC surveillance.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Jer Chen, Ph.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No